CLINICAL TRIAL: NCT01399658
Title: A Clinical Trial to Evaluate Image-Guided Gynecologic Brachytherapy in the Advanced Multimodality Image-Guided Operating Suite (AMIGO)
Brief Title: Image-Guided Gynecologic Brachytherapy
Acronym: AMIGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Martin King, MD, PhD, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-098
Record Dates: First submitted 2011-07-08; First posted 2011-07-22 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cervical Cancer; Uterine Cancer; Vaginal Cancer; Carcinoma of the Vulva
Keywords: Brachytherapy; Gynecological cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms | interventions — Brachytherapy; alovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Image-Guided Brachytherapy (Experimental): Image-guided brachytherapy
  Interventions: Procedure: Image-guided brachytherapy; Drug: 3'-Deoxy-3'-18f-Fluorothymidine

INTERVENTIONS:
Procedure: Image-guided brachytherapy — MRI-guided application of brachytherapy
  Other Names: internal radiation therapy; implant radiation
Drug: 3'-Deoxy-3'-18f-Fluorothymidine — Assessing tumor proliferation in Gynecologic cancer

SUMMARY:
Standard therapy for gynecologic cancers involves the use of brachytherapy, also called internal radiation therapy or implant radiation. The treatment being studied consists of standard brachytherapy with the additional use of MRI to guide the insertion of radioactive applicators. The purpose of the study is to find out whether MRI-guided brachytherapy is practical and beneficial when compared to the standard CT-guided brachytherapy placement. The investigators are hoping that this MRI procedure will decrease the risk of giving too high a radiation dose to the bladder or bowel.

DETAILED DESCRIPTION:
The insertion of the brachytherapy applicator will be administered in the Advanced Multimodality Image-Guided Operating (AMIGO) suite at Brigham and Women's Hospital. Subjects will undergo an MRI scan in the AMIGO suite ensuring proper placement of the applicator. Subjects may have an optional FMISO-PET scan.

Subjects will have a follow-up visit including physical exam, pap smear, and MRI of the pelvis and/or PET scan 90 days after treatment.

Subjects will have a follow-up visit including physical exam, pap smear, and MRI of the pelvis and/or PET scan 180 days after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed carcinoma of the cervix (Stage I-IVA), carcinoma of the uterus (Stage IIIB), carcinoma of the vagina (Stage I-IVA), or carcinoma of the vulva (stage I-IVA)
* Life expectancy > 6 months
* MRI of the pelvis and/or PET-CT within 4 months prior to entering study

Exclusion Criteria:

* Uncontrolled intercurrent illness
* Pacemaker, brain aneurysm clip, inner ear implant, neurostimulator, or metal fragments in the eye

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martin King, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: September 2011 to February 2016
Period: Overall Study
Arm/Group | Image-Guided Brachytherapy
Started | 93
Completed | 87
Not Completed | 6
Not completed — Ineligible | 1
Not completed — Machine Technical Issue | 3
Not completed — Alternative therapy | 1
Not completed — No reason given | 1

BASELINE CHARACTERISTICS:
Arm/Group | Image-Guided Brachytherapy
Number analyzed (Participants) | 93
Age, Continuous [Median (Full Range); unit: years] | 60 [26 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 65
  Unknown or Not Reported | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 64
  More than one race | 1
  Unknown or Not Reported | 20

OUTCOME MEASURES:

1. Primary Outcome: Mean Doses Given
Description: Doses given to the tumor, rectum, and sigmoid obtained after AMIGO-guided placement.
Time Frame: Measured while on treatment, up to 2 months.
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Image-Guided Brachytherapy
Number analyzed (Participants) | 84
Gy
  Tumor | 93.9 (8.59)
  Rectum | 63.2 (9.04)
  Sigmoid | 58.63 (12.05)

ADVERSE EVENTS:
Time Frame: From registration to 90 days post-procedure, up to 15 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Image-Guided Brachytherapy
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 86/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Image-Guided Brachytherapy (N=93)
Abdominal pain (Gastrointestinal disorders) | 21
Acidosis (Metabolism and nutrition disorders) | 2
Activated partial thrombop (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 5
Alanine aminotransferase i (Investigations) | 1
Alkaline phosphatase incre (Investigations) | 3
Alkalosis (Metabolism and nutrition disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 71
Anorexia (Metabolism and nutrition disorders) | 14
Anxiety (Psychiatric disorders) | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Aspartate aminotransferase (Investigations) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 10
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Chills (General disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 2
Cognitive disturbance (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Creatinine increased (Investigations) | 9
Cystitis noninfective (Renal and urinary disorders) | 9
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 7
Dermatitis radiation (Injury, poisoning and procedural complications) | 30
Diarrhea (Gastrointestinal disorders) | 50
Dizziness (Nervous system disorders) | 4
Duodenal hemorrhage (Gastrointestinal disorders) | 2
Dyspareunia (Reproductive system and breast disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Edema limbs (General disorders) | 4
Enterocolitis infectious (Infections and infestations) | 2
External ear inflammation (Ear and labyrinth disorders) | 1
Fatigue (General disorders) | 56
Fecal incontinence (Gastrointestinal disorders) | 1
Fever (General disorders) | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 3
Flatulence (Gastrointestinal disorders) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Generalized muscle weaknes (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 12
Hearing impaired (Ear and labyrinth disorders) | 6
Hematuria (Renal and urinary disorders) | 18
Hemorrhoids (Gastrointestinal disorders) | 10
Hot flashes (Vascular disorders) | 8
Hypercalcemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 56
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Hypocalcemia (Metabolism and nutrition disorders) | 42
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 24
Hypomagnesemia (Metabolism and nutrition disorders) | 28
Hyponatremia (Metabolism and nutrition disorders) | 28
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hypotension (Vascular disorders) | 3
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 10
Localized edema (General disorders) | 1
Lymphocyte count decreased (Investigations) | 61
Memory impairment (Nervous system disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Myositis (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 34
Neutrophil count decreased (Investigations) | 27
Pain (General disorders) | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 3
Pelvic pain (Reproductive system and breast disorders) | 16
Pelvic soft tissue necrosi (Musculoskeletal and connective tissue disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Peripheral sensory neuropa (Nervous system disorders) | 4
Platelet count decreased (Investigations) | 34
Proctitis (Gastrointestinal disorders) | 10
Proteinuria (Renal and urinary disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rectal hemorrhage (Gastrointestinal disorders) | 6
Rectal pain (Gastrointestinal disorders) | 3
Sepsis (Infections and infestations) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Stomach pain (Gastrointestinal disorders) | 1
Superficial soft tissue fi (Musculoskeletal and connective tissue disorders) | 1
Telangiectasia (Skin and subcutaneous tissue disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Urinary fistula (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 37
Urinary incontinence (Renal and urinary disorders) | 10
Urinary retention (Renal and urinary disorders) | 5
Urinary tract infection (Infections and infestations) | 7
Urinary tract obstruction (Renal and urinary disorders) | 2
Urinary tract pain (Renal and urinary disorders) | 25
Urinary urgency (Renal and urinary disorders) | 3
Urine discoloration (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 40
Vaginal dryness (Reproductive system and breast disorders) | 18
Vaginal fistula (Reproductive system and breast disorders) | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 16
Vaginal infection (Infections and infestations) | 1
Vaginal pain (Reproductive system and breast disorders) | 6
Vaginal stricture (Reproductive system and breast disorders) | 3
Vomiting (Gastrointestinal disorders) | 18
Weight gain (Investigations) | 1
Weight loss (Investigations) | 9
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
White blood cell decreased (Investigations) | 55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes